CLINICAL TRIAL: NCT05314413
Title: Examining Sex-based Differences in Metabolic and Mechanistic Responses to Disuse Induced Muscle Atrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Tyler Churchward-Venne, Principal Investigator, McGill University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: A00-M05-22B
Record Dates: First submitted 2022-03-30; First posted 2022-04-06 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Muscle Atrophy; Muscle Disuse Atrophy
Keywords: Immobilization
MeSH Terms: conditions — Muscular Atrophy; Muscular Disorders, Atrophic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single Leg Immobilization - Males (Experimental): Males will be subjected to 7-days of single-leg immobilization.
  Interventions: Procedure: Single Leg Immobilization
- Single Leg Immobilization - Females (Experimental): Females will be subjected to 7-days of single-leg immobilization.
  Interventions: Procedure: Single Leg Immobilization

INTERVENTIONS:
Procedure: Single Leg Immobilization — 7-days of single leg immobilization to induce muscle atrophy

SUMMARY:
The purpose of the proposed research is to define whether there are differences between females and males (i.e. sex-based differences) in the metabolic and mechanistic regulation of disuse-induced muscle atrophy in vivo in humans.

DETAILED DESCRIPTION:
Patients in rehabilitation may undergo periods of prolonged limb immobilization in response to injury, surgery, or illness. Due to disuse, the size and strength of muscles controlling the affected limb can decrease significantly, resulting in physical impairment or lower quality of life during the recovery phase. When measured as maximal isometric contraction, muscle strength in the immobilized limb decreases at a dramatic rate, around 1.0-1.2%/day. These declines in muscle size and strength may vary between sexes - this remains unclear. Muscle atrophy is thought to be caused by a significant decline in muscle protein synthesis (the main pathway attributing to muscle growth/ hypertrophy). There are also various pathways by which muscle is broken down. It is the sex-based differences in this muscle protein synthesis rate of decline and the pathway by which muscle is broken down that we would like to investigate for their contribution to muscle size and strength decline after a period of immobilization.

The purpose of the proposed research is to define whether there are differences between females and males (i.e. sex-based differences) in the metabolic and mechanistic regulation of disuse-induced muscle atrophy in vivo in humans.

On the participant's first visit, prior to beginning the study (Day 0), they will be instructed to fill out a health-related questionnaire, screened for all anthropometric characteristics (height, weight, age, sex) and undergo a DXA scan for body composition details. They will be familiarized with all study procedures including the muscle biopsies, strength tests, D2O, diet and exercise recording. They will also be fitted for the immobilization brace. The leg that will be immobilized will be randomized in each participant. This first visit will last approximately 2 hours. When participants return on Day 1 of the study, they will first have a lower-body MRI scan done. Following this, participants will perform single-leg strength tests on the Biodex. Thereafter on Day 2, venous blood draws and saliva samples will be taken. Participants will be administered their loading dose of D2O (5mL·kg body mass-1 of 70% D2O) and provided with daily maintenance doses of 50mL of D2O to continue to take each day for the duration of the experiment. Upon returning for Day 3, participants will undergo a single skeletal muscle biopsy from the vastus lateralis of one leg. Participants will repeat their blood and saliva sample on this day. Participants will then be outfitted with the knee brace and crutches prior to leaving the facility. Participants will also be outfitted with an ActiGraph activity monitor to record physical activity and energy expenditure while they are immobilized for 7 days. This third visit will last approximately 3 hours. Participants will monitor their own dietary intake via diet recording, which they will be instructed to carry out for 2 weekdays (i.e. Monday - Friday) and one weekend day (i.e. Saturday, Sunday). During the 7-day period of immobilization, participants will provide a saliva sample every day for measurement of 2H enrichment in body water. The saliva samples should be taken in the morning right after the participants wake up and before any food intake. Participants should drink the 1 × 50 mL maintenance dose of D2O per day provided right after collecting their saliva samples. On Day 8 participants will return to the facility to undergo post-immobilization testing which will include: a DXA scan, a lower-body MRI, two skeletal muscle biopsies (one in each leg), a blood sample, a saliva sample, and single-leg strength tests on both legs. This final visit will last approximately 4 hours.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-35 years inclusive
* Healthy, recreationally active (active for >5 hours/ week)
* Having given informed consent

Exclusion Criteria:

* Type I or Type II diabetes
* Highly trained (active for > 15 hours/week)
* Lower limb and/or back injuries in the last 6 months
* A history of thrombosis / cardiovascular disease
* Use of anticoagulants
* Musculoskeletal / orthopedic disorders
* Use of tobacco products
* Using medications known to modulate skeletal muscle metabolism including corticosteroids, hormone replacement therapy (HRT), non-steroidal anti-inflammatory drugs (i.e. paracetamol) and over-the-counter supplements including protein powder, creatine monohydrate, and fish oil
* Pregnant
* Currently participating in another clinical trial/ physical intervention research study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Fractional muscle protein synthesis rate | Integrative fractional muscle protein synthesis rates over 7 days
  Integrative fractional muscle protein synthesis rates in the immobilized and non-immobilized leg

SECONDARY OUTCOMES:
Muscle size | Baseline and 7 days
  Changes in muscle size, measured pre and post immobilization
Muscle strength | Baseline and 7 days
  Changes in muscle strength, measured pre and post immobilization
mRNA expression | Baseline and 7 days
  Changes in mRNA gene expression of specific biomarkers pertaining to skeletal muscle atrophy, measured pre and post immobilization
Protein abundance and phosphorylation | Baseline and 7 days
  Changes in protein abundance and phosphorylation status of select proteins involved in muscle protein synthesis and breakdown, measured pre and post immobilization

CONTACTS AND LOCATIONS:
Locations (1):
- Currie Gynasium 309 - McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No